CLINICAL TRIAL: NCT04194190
Title: Single Patient Protocol: A Phase II Study Using the Administration of Autologous T-Cells Genetically Engineered to Express T-Cell Receptors Reactive Against Mutated Neoantigens in a Patient With Metastatic Cancer Plus the Administration of Pembrolizumab
Brief Title: A Single Patient Will be Treated With Individual Patient TCR-Transduced PBL
Status: No longer available | Type: Expanded Access
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-C-9956; 209956 (Other: NIHCC)
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Individual Patient TCR-Transduced PBL

SUMMARY:
A single patient will be treated with Individual Patient TCR-Transduced PBL

DETAILED DESCRIPTION:
Background:

-Please refer to National Cancer Institute Surgery Branch (NCI-SB) protocol 18-C-0049, Amendment F.

Objective:

-Under Individual Patient Expanded Access, to treat a patient with metastatic breast cancer with autologous peripheral blood lymphocytes (PBL) that have been transduced with genes encoding T-cell receptors that recognize mutated neoantigens in the autologous cancer.

Eligibility:

* Must have measurable, metastatic disease as assessed per RECIST v1.1 criteria.
* Must sign the informed consent document.
* Willing to sign Durable Power of Attorney Form.
* Must have all regulatory approvals prior to start of treatment.

Design:

* Please refer to NCI-SB protocol 18-C-0049, Amendment F.
* The patient will be treated with a non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine, followed by the infusion of autologous transduced PBL and then high-dose aldesleukin. The patient will also receive pembrolizumab on Day -2 prior to cell administration and additional doses every 3 weeks following cell infusion until the time of disease progression.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult